CLINICAL TRIAL: NCT02524223
Title: Prevalence of HPV Transmission During Medically Assisted Procreation Procedures
Acronym: AMPAMAVIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1108144; 2011-A01337-34 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-13; First posted 2015-08-14 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Human Papillomavirus (HPV); Medically Assisted Procreation (MAP); Infertility
Keywords: medically assisted procreation
MeSH Terms: conditions — Infertility | interventions — Seeds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Population of couples candidate for MAP program (Other): MAP = medically assisted procreation
  Interventions: Other: Systematic HPV DNA assay in semen and cervicovaginal scrape; Other: Systematic HPV DNA cervicovaginal scrape; Other: systematic HPV Status in newborns in case of pregnancy

INTERVENTIONS:
Other: Systematic HPV DNA assay in semen and cervicovaginal scrape — Screening of HPV status at the genital level of males enrolled in MAP program.
Other: Systematic HPV DNA cervicovaginal scrape — Screening of HPV status at the genital level of females enrolled in MAP program.
Other: systematic HPV Status in newborns in case of pregnancy

SUMMARY:
Human PapillomaVirus (HPV) are ones of the main causal agents of sexually transmitted diseases. Numerous HPV genotypes such as 16, 18, 31 or 45 are considered to be at high risk of oncogenicity especially for the anal and cervical mucosa. At the present time, no recommendations exist on the risk related to HPV during Medically Assisted Procreation (MAP) procedures. The main objective of this prospective multicentric cohort study is to evaluate the prevalence of transmission of HPV via the semen during MAP program. Secondary objectives are to evaluate (1) the prevalence of HPV DNA in the sperm fractions of men enrolled in MAP, (2) the efficacy of spermatozoal pellet preparation procedures to eliminate HPV, (3) the correlation between HPV and male infertility and (4) the correlation between HPV and success rate of procreation. Results could contribute to revise guidelines of MAP procedures and HPV vaccination policy.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Age under 40 for women
* Signed informed consent by both members of the couple
* Medical indication of MAP by AI (artificial insemination), IVF(in vitro fertilization) or ICSI (intracytoplasmic sperm injection) method
* Well understanding of information letter

Exclusion Criteria:

* Age over 40 for women
* Informed consent form not signed by one or both partners
* Co-infection of one of the partners or both by HIV (human immunodeficiency virus) , HBV (hepatitis B virus) and/or HCV (hepatitis C virus)
* IVF by only frozen embryo transfer at the time of inclusion
* Severe oligospermia in male partner (<500 000 sperm cells)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 915 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2016-02-22 (Actual); Study Completion 2016-02-22 (Actual)

PRIMARY OUTCOMES:
Presence of HPV DNA on a swab sampled in the throat of newborns from one or two parents detected positive for HPV in semen and/or cervicovaginal scrape | at birth

SECONDARY OUTCOMES:
Presence of HPV DNA in seminal fractions: seminal plasma, sperm cells dedicated to MAP | At the time of enrollment, during MAP procedures and at birth (in case of)
Quantitative et qualitative parameters of spermogram analysis: volume of the ejaculate, number, mobility and morphology of sperm cells according to WHO criteria) | At the time of enrollment, during MAP procedures and at birth (in case of)
Genotype of HPV | At the time of enrollment, during MAP procedures and at birth (in case of)
Presence of HPV DNA in ovocytes samples and in embryo culture media | At the time of enrollment, during MAP procedures and at birth (in case of)
Quantitative and qualitative parameters of MAP procedures: fertilization rate, number of ovocytes, number of embryos… | At the time of enrollment, during MAP procedures and at birth (in case of)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas BOURLET, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (5):
- France (5):
  - Hôpital Jean VERDIER, Bondy
  - CHU de BORDEAUX, Bordeaux
  - CHU de CLERMONT-FERRAND, Clermont-Ferrand
  - Hôpital BICHAT, Paris
  - CHU de SAINT-ETIENNE, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No